CLINICAL TRIAL: NCT02467062
Title: Implementation of Non-size Markers Derived From 4D Flow MRI of Patients With Aortic Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Veerle Van Mossevelde, Data Nurse, Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 4D AORTIC FLOW MRI
Record Dates: First submitted 2015-06-02; First posted 2015-06-09 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Aortic Valve Disease; Aortic Aneurysm
Keywords: 4D flow
MeSH Terms: conditions — Aortic Valve Disease; Aortic Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4Dflow MRI parallel imaging (Active Comparator): 4D flow MRI with conventional parallel imaging
  Interventions: Device: MRI
- 4D flow ktARC parallel imaging (Other): 4D flow MRI kt ARC spatiotemporal parallel imaging
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — MRI measurement to evualuate for 4D blood flow pattern

SUMMARY:
The aim of the investigator is to implement 4D FLOW MRI technique into a clinical setting and evaluate the blood flow pattern and wall sheer stress in patients with aortic and/or aortic valve diseases.

DETAILED DESCRIPTION:
Currently, the timing of the replacement of the ascending aorta is solely based on the aortic diameter and concomitant valvular dysfunction and the most recent ESC guideline proposes surgical intervention of ascending aortic aneurysm in patients who have a maximal aortic diameter ≥ 55mm, regardless of etiology. On the contrary, a recent publication by Rylski et al showed that most of the dissections occur at diameters smaller than 55 mm. Several publictions have shown that the flow profile and wall sheer stress derived from 4D flow MRI are significantly different between the valve morphology, the type of the aneurysm (tubular or diffuse enlargement) and pre and postoperative patients. Clinical implementation of 4D flow may enable us to stratify the patients with aortic and/or aortic valve diseases, especially in regard to the risk of ruptures. The patients with aortic/aortic valve disease will be referred to 4D flow MRI and contrast-enhanced angiografie from the aorta clinic. Phase 1: 6 healty adult volunteers will be scanned prior to the scan of the patients and settings would be optimised for 4D flow MRI and the contrast will not be given.

Phase 2: 30 patients either scheduled for surgical treatment of their aortic disease, post-operative patients and patients under surveillance for known aortic root and/or aortic valve disease will be imaged. Only patients having a clinical indication for an MRI of the aorta/aortic valve will be included.

ELIGIBILITY:
Inclusion Criteria:

- Patients with aortic aneurysm and/or aortic valve disease older than 18 years.

Exclusion Criteria:

* Patients <18 years
* Pregnancy.
* Patients who have known contraindiction of MRI (ex claustrophobia, ICD, insulin pump etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
the bloodflow pattern | 1 day

SECONDARY OUTCOMES:
wall sheer stress | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Kaoru Tanaka, MD PhD, Principal Investigator — Department of Radiology, Universitair Ziekenhuis Brussel; Jan Nijs, MD, Principal Investigator — Brussels Center for Aortic and Cardiovascular Connective Tissue Disease
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No